CLINICAL TRIAL: NCT01442545
Title: A Study to Investigate the Effect of Multiple Doses of JNJ 39758979 on Methotrexate Pharmacokinetics in Rheumatoid Arthritis Patients on a Stable Methotrexate Dose
Brief Title: A Study to Investigate How JNJ-39758979 May Affect the Plasma Levels of Methotrexate in Rheumatoid Arthritis Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018613; 39758979ARA1001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); 2011-001227-20 (EudraCT Number)
Record Dates: First submitted 2011-08-23; First posted 2011-09-28 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; JNJ-39758979; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental)
  Interventions: Drug: JNJ-39758979 / MTX

INTERVENTIONS:
Drug: JNJ-39758979 / MTX — Day 1: MTX: Route=oral use, single dose of participant's weekly MTX dose; Days 3-15: MTX: Route=oral use, single dose of participant's weekly MTX dose and JNJ 39758979: Type=exact, unit=mg, number=300, form=tablet, route=oral use, administered daily.

SUMMARY:
The purpose of this study is to evaluate the effects of JNJ-39758979 on the pharmacokinetics (how the body handles a drug) of methotrexate in participants with rheumatoid arthritis.

DETAILED DESCRIPTION:
This is an open-label (physician and participant will know the name of the assigned drug), multi-center, non-randomized, drug-drug interaction study of JNJ-39758979 in participants with rheumatoid arthritis (RA) on a stable oral methotrexate (MTX) dose (7.5 - 25 mg). The treatment phase will last 17 days. Participants will be housed in the clinic for dosing and study procedures from Day -1 to Day 3 and again from Day 13 to Day 17. Participants completing treatment will have a follow-up visit between Days 22 and 25. Participants who discontinue the study prematurely will complete the Day 22 to 25 follow-up procedures at the time of discontinuation or as soon as possible, thereafter. The length of participation in the study for an individual participant may be up to 9 weeks (including screening). Participant safety will be monitored. Day 1: A single oral dose of the participant's weekly methotrexate dose. Days 3-15: Weekly MTX co-administered with three 100-mg, enteric-coated tablets of JNJ-39758979, administered daily.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis Functional Class I-III according to the American College of Rheumatology criteria for at least 3 months prior to Screening
* Have been treated with and tolerated oral methotrexate (taken by mouth) for a minimum of 3 months prior to screening, and must have been on a stable once-weekly methotrexate dose (taken as a single dose) between 7.5 and 25 mg/week for a minimum of 1 month prior to Day 1
* Participants may continue on stable nonsteroidal anti-inflammatory drug (NSAID) and/or corticosteroid background therapy for rheumatoid arthritis (RA) or stable therapies for other conditions as prescribed by physician, providing that the doses of such therapy are stable for at least 1 month prior to screening and will remain unchanged for the entire study duration
* Medically stable on the basis of physical examination, medical history, vital signs, and electrocardiogram (ECG) performed at screening
* Laboratory values within certain limits at screening and Day-1. Abnormalities consistent with those observed in patients with RA are permissible.

Exclusion Criteria:

* History of or current clinically significant medical illness as specified on the protocol, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Have been treated with a monoclonal antibody for RA in the 3 months prior to enrollment or have had a serious infection within 2 weeks of the study treatment period
* Except for methotrexate, treated with approved or investigational non-biologic disease-modifying antirheumatic drugs (DMARDs) during the 4 weeks or 5 half-lives prior to the first dose of JNJ-39758979, whichever is longer. These agents include, but are not limited to D-penicillamine, hydroxychloroquine, chloroquine, oral or parenteral gold salts, sulfasalazine, leflunomide, azathioprine, cyclosporine, tacrolimus and mycophenolate mofetil.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-08; Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Blood levels of methotrexate | Up to approximately 7 weeks
  To assess the effect of multiple doses of JNJ-39758979 on blood levels of methotrexate

SECONDARY OUTCOMES:
Blood levels of JNJ 39758979 | Up to approximately 7 weeks
  To assess the effect of MTX on the blood levels of JNJ 39758979
The number of participants with adverse events | Up to approximately 7 weeks
Clinical laboratory tests | Up to approximately 7 weeks
  Blood and urine tests
Electrocardiograms | Up to approximately 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: J&J Pharmaceutical Research & Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (5):
- United States (3):
  - Daytona Beach, Florida
  - Duncansville, Pennsylvania
  - Dallas, Texas
- Germany (2):
  - Berlin
  - Munich